# **Protocol**

# ECHO study

# The Effect of Copper on the Healing of Obstetric wounds VERSION 3 - 17/09/2015

#### Authors:

L.P. Arendsen MD, Research Fellow in Urogynaecology

R. Thakar MD, FRCOG, Consultant Obstetrician & Gynaecologist, Urogynaecology subspecialist

A.H. Sultan MD, FRCOG, Consultant Obstetrician & Gynaecologist

Croydon University Hospital

530 London Road, CR7 7YE

Croydon, United Kingdom

Telephone number: 020 8401 3000

**Full title:** Randomised controlled trial on the effect of copper impregnated dressings and maternity pads on the healing of obstetric wounds and wound infection

#### Background

In Croydon Health Services around 4,000 babies are born annually and the vast majority are born vaginally. The most common complication of vaginal delivery is perineal or vaginal laceration with a prevalence as high as 85% and up to 70% will need suturing (1). Within Croydon Health Services 73% deliver vaginally of whom 66% sustain perineal laceration (19% first degree, 74% second degree, 7% 3<sup>rd</sup>/4<sup>th</sup> degree) and an episiotomy is performed in 24% of the vaginal deliveries. Minor lacerations are often left unsutured, whereas the majority of the second or higher degree tears will be sutured directly after delivery. Due to supporting factors such as a moist environment and the presence of high numbers of bacteria, perineal trauma is associated with wound infection and affects 11% of the women with sutured tears (2). Wound infection can cause pain, dehiscence, delayed wound healing and interfere with a woman's ability to nurture their baby and enjoy motherhood (3).

The caesarean section rate worldwide is rising (4) and the rate in Croydon University

Hospital is in the region of 25% of all deliveries. The most significant source of maternal
morbidity after caesarean section is postoperative infection (surgical site infection) and can
be the cause of a prolonged hospital stay, readmissions (5) sepsis and maternal death (6).

Surgical site infection is one of the most prevalent reported nosocomial infection, which
accounts for 14-16% of all hospital-acquired infections. Despite prophylactic antibiotics, the
rate of wound infection after caesarean section is ranging between 7% and 41% (7-9).

According to the Centers for Disease Control and Prevention (CDC), surgical site infection
can be classified as an incisional infection, either superficial or deep, or an organ or space
infection, such as endometritis (10). See figure one for the CDC surgical site classification.

Figure 1 CDC Classification for Surgical Site Infections



The micro-organisms that are most commonly the cause of the infection of perineal tears and caesarean section wounds are Enterococci, Streptococci, Staphylococci, Gram-negative bacteria and anaerobes (5, 11). As a consequence of antibiotic resistance, MRSA infection is becoming an increasing challenge. Several studies have detected MRSA colonisation rates of up to 10% in rectovaginal swabs in asymptomatic pregnant women (12, 13). MRSA has been proven to cause more severe postpartum infections, especially after caesarean section (14-16). Although several strategies to eliminate or reduce colonisation of MRSA such as skin wash have been studied, the real efficacy of such interventions remains inconclusive (17). Moreover, the preoperative skin preparation using chlorhexidine, which reduced the overall rate of surgical site infection, was found ineffective among MRSA carriers (18).

#### Antimicrobial copper

The antimicrobial effect of copper has been known for centuries. As early as 2600-2200 BC the Egyptians used green copper rust for the treatment of chest wounds and to sterilise drinking water. In another Papyrus it was written that copper splinters, shavings and various

copper salts and oxides were used to treat headaches, burn wounds, itching and skin infections (19). With the increase in antibiotic resistant bacteria causing nosocomial infections, copper has become a popular subject of recent research. There are many laboratory studies showing the biocidal effect of copper on a wide range of microbes such as bacteria, fungi and viruses (20, 21). Copper has also been proven to be effective against Methicillin-resistant Staphylococcus aureus (MRSA) (22) and Vancomycin-resistant Enterococci (VRE) (23). The use of copper surfaces within the hospital setting has been evaluated in several clinical studies showing significant reductions in bacterial colonisation on copper surfaces compared to standard materials (24). After the use of copper as a biocidal contact surface, the use of copper impregnated textiles was explored. Although there is a variety of containing copper impregnated textiles available such as socks, pyjamas, underwear, bed linen, face masks, stockings and wound dressings, there is a paucity of clinical research. There has however been a clinical study on the effect of copper impregnated socks in patients suffering from tinea pedis and this revealed a significant improvement or resolution of the infection after wearing these socks for two weeks (25).

#### Wound healing

Copper is assumed to be involved in several processes crucial for wound healing (26). A key role in wound healing is angiogenesis. It has been shown that copper induces the production of vascular endothelial growth factor (VEGF) and therefore stimulates angiogenesis (27). Furthermore, copper promotes wound healing due to an elevation in integrin expression (28); enhancement of fibrinogen stabilisation (29) and up regulation of several enzymes essential for matrix remodelling and cell growth (30). Several laboratory studies have demonstrated an association between a copper dependant enzyme, lysyl oxidase (LOX), and skin ageing and pathological skin conditions (31).

## Safety

The dermal exposure to copper is considered safe as copper is not only an essential element for normal skin function but also essential for the immune system and blood coagulation (32). In contrast to microorganisms, human skin cells have the ability to metabolise and utilise copper (33) and therefore the development of adverse reactions are unlikely.

Our hypothesis is that copper impregnated fibres in maternity pads and surgical wound dressings, reduces infection rates in perineal lacerations, episiotomies and caesarean section wounds.

## Aim

The aim of this study is to investigate the impact of copper impregnated wound dressings and maternity pads on the incidence of infection in perineal wounds after vaginal delivery and caesarean section wounds.

## **Objectives**

## Primary:

- To assess the effect of copper impregnated wound dressings on the incidence of wound infection following caesarean section.
- 2. To assess the effect of copper impregnated maternity pads on the incidence of wound infection of second degree perineal tears following vaginal delivery.

## Secondary:

- 1. To assess the effect of copper impregnated wound dressings on other maternal outcomes, such as length of hospitalisation, readmission rate and pain of the wound.
- 2. To assess the effect of copper impregnated maternity pads on other maternal outcomes, such as length of hospitalisation, readmission rate and perineal pain.

## Methodology

This is a double blind randomised controlled pilot study to assess feasibility of copper impregnated wound dressings and maternity pads for the healing of obstetric wounds. All pregnant women in Croydon University Hospital who attend their routine second-trimester scan appointment at approximately 20 weeks of gestation will receive a detailed patient information sheet (Appendix 1 Patient Information Sheet) about the four arms of this study. When women are eligible to participate after delivery, informed consent will be obtained (see Appendix 2 Informed Consent).

All women who are planned to have an elective caesarean section will be recruited at their antenatal clinic appointment. A detailed patient information sheet specific for the caesarean section arm of this study will be given prior to consent. Informed consent will be obtained antenatally. After caesarean section, confirmation of willingness to participate in this study will be obtained and documented directly after elective caesarean.

All patients will be assessed by telephone at baseline, 7, 14, and 30 days. The recruitment period will be 12 months.

#### The inclusion criteria are:

- Aged 18 or over
- Delivered by caesarean section (emergency or elective),
   or vaginally, sustaining a perineal tear or episiotomy which needed to be sutured
- Ability to understand the content of the patient information sheet (in English, via an interpreter if needed and possible)
- Ability to give informed consent

#### The exclusion criteria are:

- Inability to give consent
- Fetal or neonatal death or poor neonatal outcome
- Obstetric anal sphincter injuries
- Included in another study on postpartum infection conducted in the Obstetrics and Gynaecology Department
- Wilson's disease
- Allergy to copper

#### Randomisation

After inclusion all patients will be randomised for a wound dressing or maternity pad with (study group) or without copper (control group). The two sets of wound dressings and pads will be marked "A" or "B". Both the clinician and the patient will be blinded to the randomised group. Only the manufacturer will be aware of which group contains copper.

#### Copper impregnated dressings

As soon as possible, but within 12 hours after primary closure of the caesarean section incision, the randomised study dressing will be applied. The two study dressings will be equivalent to the dressing normally used within this Trust, except that one set of dressings will have a thin top layer of non-woven polyester fibres with 3% copper oxide ions permanently attached to it. According to local protocol the wound dressing will be left intact for 7 days following surgery and will be renewed if necessary.

#### Copper impregnated maternity pads

As soon as possible, but within 12 hours after suturing women will be asked to wear the study maternity pads, which will be provided. The two sets of study maternity pads will be equivalent to the currently recommended pads, except that one set of pads will have a thin

top layer of non-woven polyester fibres with 3% copper oxide ions permanently attached to it. Women will be asked to use the pads for 14 days after delivery.

### Patient data, history and physical examination:

Demographic data such as age, ethnicity, height and weight will be collected as well as obstetric data and delivery details (Appendix 4 Datasheet). Past medical history such as concomitant (chronic) diseases and the use of medications will be obtained. Wound infection will be assessed via a telephone questionnaire after 7, 14 and 30 days after delivery.

The data will be stored in a secure room within Trust facilities. All electronic data will be stored within password protected IT system within the Trust, which is only accessible by the clinical and research team.

## Questionnaire

For the assessment of surgical site infection, the Post Discharge Questionnaire (see Appendix 5 Post Discharge Questionnaire) used by the HPC surgical site infection surveillance will be used, which is according to the worldwide used definition of surgical site infection by the CDC (10). Since the Post Discharge Questionnaire is dependent on the women's report rather than confirmation following clinical assessment of the wound, the criteria for infection have modified to allow for easy interpretation of the reported symptoms as follows:

- Criterion 1: discharge pus AND antibiotics prescribed
- Criterion 2: clinical signs\* AND dehiscence
- Criterion 3: Clinical signs\* AND antibiotics prescribed
   \*clinical signs: at least 2 of the following must be present: pain, heat, redness or swelling

Without clinical assessment of the wound, the type of SSI cannot be defined.

Since there is no commonly used definition in the literature for wound infection following perineal tears, the Post discharge Questionnaire with the modified criteria for infection will be used for the perineal tears as well.

## Microbiological assessment

When wound infection is suspected according to the above explained criteria, a wound swab is taken to detect the causative organisms.

## Statistical analysis

Statistical analysis will be performed using SPSS version 20.0 or higher. Infection rates in the perineal tear group and the caesarean section group will be analysed. The infection rates in the study group (with copper) will be compared to the control group and possible risk factors for infection will be explored.

## Sample size calculation

Since the effect of copper on infection rates is currently unknown, we will conduct a pilot study for 12 months. After 3 months we will perform an interim analysis to be able to calculate the sample size.

| Maternity statistics at Croydon University Hospital | |
|------------------------------------------------------|----------------|
| | Past 12 months |
| | (N=3752) |
| Vaginal deliveries (N=2734) | |
| Episiotomy | 643 |
| 2nd degree tear | 1334 |
| Total sutured tears | 1977 |
| (excl 3 <sup>rd</sup> /4 <sup>th</sup> degree tears) | |
| Caesarean Section (N=1018) | |
| EmCS | 696 |
| EICS | 322 |
| Total study population | 2995 |

#### References

- 1. McCandlish, R,Bowler, U,van Asten, H,Berridge, G,Winter, C,Sames, L,Garcia, J,Renfrew, M,Elbourne, D. A randomised controlled trial of care of the perineum during second stage of normal labour. British journal of obstetrics and gynaecology, vol. 105, no. 12, p. 1262-1272, 0306-5456 (December 1998)
- 2. Johnson, Adeyemi, Thakar, Ranee, Sultan, Abdul H. Obstetric perineal wound infection: is there underreporting? British journal of nursing (Mark Allen Publishing), vol. 21, no. 5, p. S28, 0966-0461 (2012 Mar 8-21)
- American College of Obstetrics and Gynecology. Operative vaginal delivery. Clinical management guidelines for obstetrician-gynecologists. American College of Obstetrics and Gynecology. International journal of gynaecology and obstetrics: the official organ of the International Federation of Gynaecology and Obstetrics, vol. 74, no. 1, p. 69-76, 0020-7292 (July 2001)
- 4. Thomas, J,Callwood, A,Brocklehurst, P,Walker, J. The National Sentinel Caesarean Section Audit. BJOG: an international journal of obstetrics and gynaecology, vol. 107, no. 5, p. 579-580, 1470-0328 (May 2000)
- 5. Smaill, Fiona M,Grivell, Rosalie M. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. The Cochrane database of systematic reviews, vol. 10, p. CD007482. (2014)
- Declercq, Eugene, Barger, Mary, Cabral, Howard J, Evans, Stephen R, Kotelchuck, Milton, Simon, Carol, Weiss, Judith, Heffner, Linda J. Maternal outcomes associated with planned primary cesarean births compared with planned vaginal births.
   Obstetrics and gynecology, vol. 109, no. 3, p. 669-677, 0029-7844 (March 2007)
- 7. Hillan EM. Postoperative morbidity following Caesarean delivery. J Adv Nurs 1995;22:1035e1042.
- 8. Henderson E, Love EJ. Incidence of hospital-acquired infections associated with caesarean section. J Hosp Infect 1995; 29:245e255.
- Ward, V P, Charlett, A, Fagan, J, Crawshaw, S C. Enhanced surgical site infection surveillance following caesarean section: experience of a multicentre collaborative post-discharge system. The Journal of hospital infection, vol. 70, no. 2, p. 166-173, 0195-6701 (October 2008)
- Mangram, A J,Horan, T C,Pearson, M L,Silver, L C,Jarvis, W R. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infection control and hospital epidemiology, vol. 20, no. 4, p. 250, 0899-823X (April 1999)
- 11. Martens MG, Kolrud BL, Faro S, Maccato M, Hammill H. Development of wound infection or separation after cesarean delivery. Prospective evaluation of 2,431 cases. *Journal of Reproductive Medicine* 1995;40:171–5.

- 12. Creech, C Buddy,Litzner, Brandon,Talbot, Thomas R,Schaffner, William. Frequency of detection of methicillin-resistant Staphylococcus aureus from rectovaginal swabs in pregnant women. American journal of infection control, vol. 38, no. 1, p. 72-74 (February 2010)
- 13. Beigi, R,Hanrahan, J. Staphylococcus aureus and MRSA colonization rates among gravidas admitted to labor and delivery: a pilot study. Infectious diseases in obstetrics and gynecology, vol. 2007, p. 70876. (2007)
- Stumpf, Paul G,Flores, Marisol, Murillo, Jeremias. Serious postpartum infection due to MRSA in an asymptomatic carrier: case report and review. American journal of perinatology, vol. 25, no. 7, p. 413-415 (August 2008)
- 15. Thurman AR, Anca Y, White CA, Soper DE. Postcesarean delivery infectious morbidity: Focus on preoperative antibiotics and methicillin-resistant Staphylococcus aureus. Am J Infect Control 2010;38:612–6.
- American College of Obstetricians and Gynecologists. ACOG Practice Bulletin No.
   120: Use of prophylactic antibiotics in labor and delivery. Obstetrics and gynecology,
   vol. 117, no. 6, p. 1472-1483 (June 2011)
- 17. Liu C, Bayer A, Cosgrove SE, et al. Clinical practice guidelines by the Infectious Diseases Society of America for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis 2011;52:1–38.
- Whitman TJ, Herlihy RK, Schlett CD, et al. Chlorhexidineimpregnated cloths to prevent skin and soft-tissue infection in marine recruits: a cluster-randomized, double- blind, controlled effectiveness trial. Infect Control Hosp Epidemiol 2010;12:1207–15.
- 19. Dollwet HHA, Sorenson JRJ. Historic uses of copper compounds in medicine. Trace Elements Med 1985; 2: 80-7.
- 20. Borkow G, Gabbay J. Copper as a biocidal tool. *Curr Med Chem* 2005; 12: 2163-2175
- 21. Borkow G, Gabbay J. Copper, an ancient remedy returning to fight microbial, fungal and viral infections. *Curr Chem Biol* 2009; 3: 272-278
- 22. Noyce JO, Michels H, Keevil CW. Potential use of copper surfaces to reduce survival of epidemic meticillin-resistant Staphylococcus aureus in the healthcare environment. J Hosp Infect 2006;63:289e297.
- 23. Warnes SL, Keevil CW. Mechanism of copper surface toxicity in vancomycin-resistant enterococci following wet or dry surface contact. Appl Environ Microbiol 2011;77:6049e6059.
- 24. O'Gorman J, Humphreys H, Application of copper to prevent and control infection. Where are we now? Journal of Hospital Infection (2012), hhtp://dx.doi.org/10.1016/j.jhin.2012.05.009

- 25. Gargiulo, ME., Del Carmen-Elias, A. And Borkow, G. Analysis of the effect of wearing copper oxide impregnated socks on *tinea pedis* based on "before and after" pictures a statistical follow-up tool. *The Open Biology Journal*, 2012, vol. 5, no. p. 17-22.
- 26. Borkow G, Gabbay J, Zatcoff RC. Could chronic wounds not heal due to too low local copper levels? Med Hypotheses 2008; 70: 610–3.
- 27. Sen CK, Khanna S, Venojarvi M, Trikha P, Ellison EC, Hunt TK, Roy S. Copper-induced vascular endothelial growth factor expression and wound healing. Am J Physiol Heart Circ Physiol 2002; 282: H1821–7.
- 28. Tenaud I, Sainte-Marie I, Jumbou O, Litoux P, Dreno B. In vitro modulation of keratinocyte wound healing integrins by zinc, copper and manganese. Br J Dermatol 1999; 140: 26–34.
- 29. Ahmed Z, Briden A, Hall S, Brown RA. Stabilisation of cables of fibronectin with micromolar concentrations of copper: in vitro cell substrate properties. Biomaterials 2004; 25: 803–12.
- 30. Rucker RB, Kosonen T, Clegg MS, Mitchell AE, Rucker BR, Uriu-Hare JY, Keen CL. Copper, lysyl oxidase, and extracellular matrix protein cross-linking. Am J Clin Nutr 1998; 67: 996S–1002S.
- 31. Szauter KM, Cao T, Boyd CD, Csiszar K. Lysyl oxidase in development, aging and pathologies of the skin. Pathol Biol (Paris) 2005;53:448–56.
- 32. Uauy R, Olivares M, Gonzalez M. Essentiality of copper in humans. Am J Clin Nutr 1998; 67: 952S–9S.
- 33. Hostynek JJ, Dreher F, Maibach HI. Human skin penetration of a copper tripeptide in vitro as a function of skin layer. Inflammation Research, 01 2011, vol./is. 60/1(79-86), 1023-3830;1420-908X (2011 Jan)